CLINICAL TRIAL: NCT01732627
Title: Immunogenicity and Safety of a Quadrivalent Meningococcal Conjugate Vaccine Administered in Subjects 56 Years of Age and Older
Brief Title: Study of a Quadrivalent Meningococcal Conjugate Vaccine in Subjects Aged 56 and Older
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MET44; U1111-1127-6804 (Other: WHO)
Record Dates: First submitted 2012-11-13; First posted 2012-11-26 (Estimated); Results first posted 2020-06-09 (Actual); Last update posted 2022-04-04 (Actual); Status verified 2022-03

CONDITIONS: Meningitis; Meningococcal Meningitis; Meningococcal Infections; Invasive Meningococcal Disease
Keywords: Meningitis; Meningococcal Meningitis; Menactra®; Menomune® A/C/Y/W 135
MeSH Terms: conditions — Meningitis; Meningitis, Meningococcal; Meningococcal Infections | interventions — Meningococcal Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group 1: MenACYW Conjugate Vaccine (Experimental): Adult participants aged greater than or equal to (≥) 56 years received a single dose of Meningococcal Polysaccharide (Serogroups A, C, Y, and W 135) Tetanus Toxoid (MenACYW) Conjugate vaccine on Day 0.
  Interventions: Biological: Meningococcal Polysaccharide (A, C, Y, and W 135) Tetanus Protein Conjugate Vaccine
- Group 2: Menomune® A/C/Y/W 135 vaccine (Active Comparator): Adult participants aged ≥56 years received a single dose of Meningococcal Polysaccharide Vaccine, Groups A, C, Y, and W 135 Combined (Menomune®) vaccine on Day 0.
  Interventions: Biological: Meningococcal Polysaccharide Vaccine, Groups A, C, Y, W 135 Combined

INTERVENTIONS:
Biological: Meningococcal Polysaccharide (A, C, Y, and W 135) Tetanus Protein Conjugate Vaccine — 0.5 milliliter (mL), Intramuscular (IM)
  Other Names: MenACYW Conjugate Vaccine
  Arms: Group 1: MenACYW Conjugate Vaccine
Biological: Meningococcal Polysaccharide Vaccine, Groups A, C, Y, W 135 Combined — 0.5 mL, Subcutaneous (SC)
  Other Names: Menomune® A/C/Y/W 135
  Arms: Group 2: Menomune® A/C/Y/W 135 vaccine

SUMMARY:
Primary objectives:

* To describe the antibody responses to meningococcal serogroups A, C, Y, and W 135, measured by serum bactericidal assay using human complement (hSBA) and baby rabbit complement (rSBA), induced by a single dose of Meningococcal Polysaccharide (A, C, Y, and W 135) Tetanus Protein (MenACYW) Conjugate vaccine or Menomune® - A/C/Y/W 135.
* To describe the safety profile of a single dose of MenACYW Conjugate vaccine or Menomune® - A/C/Y/W 135.

DETAILED DESCRIPTION:
All participants received a single dose of their assigned vaccine on Day 0. They were assessed for immunogenicity on Day 0 and Day 30, and monitored for safety throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Aged 56 or older on the day of inclusion.
* Informed consent form had been signed and dated.
* Able to attend all scheduled visits and complied with all trial procedures.

Exclusion Criteria:

* Participant was pregnant, or lactating, or of childbearing potential (were considered of non-childbearing potential, a female must be post-menopausal for at least 1 year, surgically sterile, or used an effective method of contraception or abstinence from at least 4 weeks prior to vaccination and until at least 4 weeks after vaccination).
* Participation at the time of study enrollment (or in the 4 weeks preceding the trial vaccination) or planned participation during the present trial period in another clinical trial investigating a vaccine, drug, medical device, or medical procedure.
* Receipt of any vaccine in the 4 weeks preceding the trial vaccination or planned receipt of any vaccine in the 4 weeks following the trial vaccination except for influenza vaccination, which might be received at least 2 weeks before or after the study vaccines.
* Previous vaccination against meningococcal disease with either a trial vaccine or another vaccine.
* Receipt of immune globulins, blood or blood-derived products in the past 3 months.
* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy, such as anti-cancer chemotherapy or radiation therapy, within the preceding 6 months; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months).
* History of meningococcal infection, confirmed either clinically, serologically, or microbiologically.
* At high risk for meningococcal infection during the trial.
* Known systemic hypersensitivity to latex or any of the vaccine components, or history of a severe reaction to the vaccines used in the trial or to a vaccine containing any of the same substances.
* Personal history of Guillain-Barré syndrome.
* Personal history of an Arthus-like reaction after vaccination with a tetanus toxoid-containing vaccine within at least 10 years of the proposed study vaccination.
* Self-reported thrombocytopenia, contraindicating IM vaccination.
* Bleeding disorder, or receipt of anticoagulants in the 3 weeks preceding inclusion, contraindicating IM vaccination.
* Deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized involuntarily.
* Current alcohol abuse or drug addiction.
* Chronic illness that, in the opinion of the investigator, was at a stage where it might interfere with trial conduct or completion.
* Moderate or severe acute illness/infection (according to investigator judgment) on the day of vaccination or febrile illness (temperature ≥ 100.4°Fahrenheit [≥ 38.0°Celsius]). A prospective participant should not be included in the study until the condition had resolved or the febrile event had subsided.
* Receipt of oral or injectable antibiotic therapy within 3 days prior to any blood draw. Should a participant receive oral or injectable antibiotic therapy within 3 days prior to any blood draw, the Investigator would postpone the blood draw until it had been 3 days since the participant last received oral or injectable antibiotic therapy. Postponement must still be within the timeframe for blood draw indicated in the Table of Study Procedures, when possible.
* Identified as an Investigator or employee of the Investigator or study center with direct involvement in the proposed study, or identified as an immediate family member (i.e., parent, spouse, natural or adopted child) of the Investigator or employee with direct involvement in the proposed study.

Min Age: 56 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 301 (Actual)
Dates: Start 2012-11-12 (Actual); Primary Completion 2013-01-17 (Actual); Study Completion 2013-01-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur Inc.
Locations (12):
- United States (12):
  - Chandler, Arizona
  - Scottsdale, Arizona
  - Denver, Colorado
  - Milford, Connecticut
  - Edina, Minnesota
  - St Louis, Missouri
  - Columbus, Ohio
  - Anderson, South Carolina
  - Murray, Utah
  - Salt Lake City, Utah
  - West Jordan, Utah
  - Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Result] Kirstein J, Pina M, Pan J, Jordanov E, Dhingra MS. Immunogenicity and safety of a quadrivalent meningococcal tetanus toxoid-conjugate vaccine (MenACYW-TT) in adults 56 years of age and older: a Phase II randomized study. Hum Vaccin Immunother. 2020 Jun 2;16(6):1299-1305. doi: 10.1080/21645515.2020.1733868. Epub 2020 Apr 1. PMID 32233961

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was conducted from 12-November-2012 to 17-January-2013 at 12 sites in the United States.
Pre-assignment Details: A total of 301 participants were enrolled and vaccinated in the study.
Period: Overall Study
Arm/Group | Group 1: MenACYW Conjugate Vaccine | Group 2: Menomune® A/C/Y/W 135 Vaccine
Started (Randomized and vaccinated.) | 201 | 100
Safety Analysis Set (SafAS) (Participants who received at least 1 dose of study or control vaccine and had safety data available.) | 199 | 100
Completed | 200 | 100
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: Analysis was performed on all randomized participants.
Groups:
- Group 1: MenACYW Conjugate Vaccine: Adult participants aged ≥56 years received a single dose of MenACYW Conjugate vaccine on Day 0.
- Group 2: Menomune® A/C/Y/W 135 Vaccine: Adult participants aged ≥56 years received a single dose of Menomune® vaccine on Day 0.
- Total: Total of all reporting groups
Arm/Group | Group 1: MenACYW Conjugate Vaccine | Group 2: Menomune® A/C/Y/W 135 Vaccine | Total
Number analyzed (Participants) | 201 | 100 | 301
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.0 (7.15) | 65.8 (6.58) | 65.9 (6.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 121 | 55 | 176
  Male | 80 | 45 | 125
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 2 | 9
  White | 190 | 97 | 287
  More than one race | 3 | 1 | 4
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Antibody Titers ≥1:4 and ≥1:8 Measured by Serum Bactericidal Assay Using Human Complement (hSBA) Against Meningococcal Serogroups A, C, Y, and W 135 Before Vaccination With MenACYW Conjugate Vaccine or Menomune® Vaccine
Description: Antibody titers against meningococcal serogroups A, C, Y, and W 135 were measured by hSBA assay method.
Time Frame: Day 0 (pre-vaccination)
Population: Analysis was performed on Per-Protocol Analysis Set (PPAS) population which included participants who received at least one dose of the study vaccine, had any valid serology result, and no protocol deviations.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: MenACYW Conjugate Vaccine | Group 2: Menomune® A/C/Y/W 135 Vaccine
Number analyzed (Participants) | 195 | 94
percentage of participants
  Serogroup A: ≥1:4 | 95.9 [92.1 to 98.2] | 96.8 [91.0 to 99.3]
  Serogroup A: ≥1:8 | 76.4 [69.8 to 82.2] | 79.8 [70.2 to 87.4]
  Serogroup C: ≥1:4 | 27.7 [21.5 to 34.5] | 30.9 [21.7 to 41.2]
  Serogroup C: ≥1:8 | 17.4 [12.4 to 23.5] | 10.6 [5.2 to 18.7]
  Serogroup Y: ≥1:4 | 22.1 [16.4 to 28.5] | 26.6 [18.0 to 36.7]
  Serogroup Y: ≥1:8 | 13.3 [8.9 to 18.9] | 24.5 [16.2 to 34.4]
  Serogroup W 135: ≥1:4 | 26.2 [20.1 to 32.9] | 26.6 [18.0 to 36.7]
  Serogroup W 135: ≥1:8 | 13.3 [8.9 to 18.9] | 8.5 [3.7 to 16.1]

2. Primary Outcome: Percentage of Participants With Antibody Titers ≥1:4 and ≥1:8 Measured by hSBA Against Meningococcal Serogroups A, C, Y, and W 135 Following Vaccination With MenACYW Conjugate Vaccine or Menomune® Vaccine
Description: Antibody titers against meningococcal serogroups A, C, Y, and W 135 were measured by hSBA assay method.
Time Frame: Day 30 (post-vaccination)
Population: Analysis was performed on PPAS population.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: MenACYW Conjugate Vaccine | Group 2: Menomune® A/C/Y/W 135 Vaccine
Number analyzed (Participants) | 195 | 94
percentage of participants
  Serogroup A: ≥1:4 | 97.4 [94.1 to 99.2] | 93.6 [86.6 to 97.6]
  Serogroup A: ≥1:8 | 93.8 [89.5 to 96.8] | 85.1 [76.3 to 91.6]
  Serogroup C: ≥1:4 | 85.6 [79.9 to 90.2] | 79.8 [70.2 to 87.4]
  Serogroup C: ≥1:8 | 74.9 [68.2 to 80.8] | 62.8 [52.2 to 72.5]
  Serogroup Y: ≥1:4 | 87.2 [81.7 to 91.5] | 73.4 [63.3 to 82.0]
  Serogroup Y: ≥1:8 | 80.5 [74.2 to 85.8] | 59.6 [49.0 to 69.6]
  Serogroup W 135: ≥1:4 | 88.7 [83.4 to 92.8] | 77.7 [67.9 to 85.6]
  Serogroup W 135: ≥1:8 | 79.5 [73.1 to 84.9] | 60.6 [50.0 to 70.6]

3. Primary Outcome: Percentage of Participants With Vaccine Seroresponse Measured by hSBA Against Meningococcal Serogroups A, C, Y, and W 135 Following Vaccination With MenACYW Conjugate Vaccine or Menomune® Vaccine
Description: Vaccine seroresponse for serogroups A, C, Y, and W 135 was measured by hSBA assay method. Seroresponse was defined as post-vaccination hSBA titers ≥1:8 for participants with pre-vaccination hSBA titers less than (<) 1:8, or at least a 4-fold increase in hSBA titers from pre- to post-vaccination for participants with pre-vaccination hSBA titers ≥1:8.
Time Frame: Day 30 (post-vaccination)
Population: Analysis was performed on PPAS population.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: MenACYW Conjugate Vaccine | Group 2: Menomune® A/C/Y/W 135 Vaccine
Number analyzed (Participants) | 195 | 94
percentage of participants
  Serogroup A | 65.1 [58.0 to 71.8] | 46.8 [36.4 to 57.4]
  Serogroup C | 70.8 [63.8 to 77.0] | 59.6 [49.0 to 69.6]
  Serogroup Y | 75.4 [68.7 to 81.3] | 48.9 [38.5 to 59.5]
  Serogroup W 135 | 74.4 [67.6 to 80.3] | 55.3 [44.7 to 65.6]

4. Primary Outcome: Geometric Mean Titers (GMTs) of Antibodies Against Meningococcal Serogroups A, C, Y, and W 135 Measured by hSBA Before Vaccination With MenACYW Conjugate Vaccine or Menomune® Vaccine
Description: GMTs of antibodies against meningococcal serogroups A, C, Y, and W 135 were measured by hSBA assay method.
Time Frame: Day 0 (pre-vaccination)
Population: Analysis was performed on PPAS population.
Measure: Geometric Mean (95% Confidence Interval); unit: titers (1/dilution)
Arm/Group | Group 1: MenACYW Conjugate Vaccine | Group 2: Menomune® A/C/Y/W 135 Vaccine
Number analyzed (Participants) | 195 | 94
titers (1/dilution)
  Serogroup A | 9.73 [8.65 to 10.9] | 10.4 [8.58 to 12.5]
  Serogroup C | 3.32 [2.87 to 3.85] | 2.87 [2.49 to 3.31]
  Serogroup Y | 3.02 [2.63 to 3.47] | 3.53 [2.84 to 4.38]
  Serogroup W 135 | 2.83 [2.56 to 3.14] | 2.83 [2.40 to 3.33]

5. Primary Outcome: Geometric Mean Titers (GMTs) of Antibodies Against Meningococcal Serogroups A, C, Y, and W 135 Measured by hSBA Following Vaccination With MenACYW Conjugate Vaccine or Menomune® Vaccine
Description: GMTs of antibodies against meningococcal serogroups A, C, Y, and W 135 were measured by hSBA assay method.
Time Frame: Day 30 (post-vaccination)
Population: Analysis was performed on PPAS population.
Measure: Geometric Mean (95% Confidence Interval); unit: titers (1/dilution)
Arm/Group | Group 1: MenACYW Conjugate Vaccine | Group 2: Menomune® A/C/Y/W 135 Vaccine
Number analyzed (Participants) | 195 | 94
titers (1/dilution)
  Serogroup A | 51.0 [40.7 to 63.9] | 31.8 [22.5 to 44.9]
  Serogroup C | 48.3 [34.8 to 67.1] | 18.5 [12.1 to 28.3]
  Serogroup Y | 41.9 [31.8 to 55.3] | 16.6 [11.3 to 24.5]
  Serogroup W 135 | 29.0 [22.5 to 37.3] | 17.1 [11.6 to 25.2]

6. Primary Outcome: Percentage of Participants With Antibody Titers ≥1:8 and ≥1:128 Measured by Serum Bactericidal Assay Using Baby Rabbit Complement (rSBA) Against Meningococcal Serogroups A, C, Y, and W 135 Before Vaccination With MenACYW Conjugate Vaccine or Menomune®
Description: Antibody titers against meningococcal serogroups A, C, Y, and W 135 were measured by rSBA assay method.
Time Frame: Day 0 (pre-vaccination)
Population: Analysis was performed on PPAS population. Here, 'Number analyzed' = participants with available data for each specified category.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: MenACYW Conjugate Vaccine | Group 2: Menomune® A/C/Y/W 135 Vaccine
Number analyzed (Participants) | 195 | 94
percentage of participants
  Serogroup A: ≥1:8: number analyzed (Participants) | 195 | 93
  Serogroup A: ≥1:8 | 28.2 [22.0 to 35.1] | 26.9 [18.2 to 37.1]
  Serogroup A: ≥1:128: number analyzed (Participants) | 195 | 93
  Serogroup A: ≥1:128 | 22.1 [16.4 to 28.5] | 22.6 [14.6 to 32.4]
  Serogroup C: ≥1:8 | 12.3 [8.0 to 17.8] | 9.6 [4.5 to 17.4]
  Serogroup C: ≥1:128 | 8.2 [4.8 to 13.0] | 4.3 [1.2 to 10.5]
  Serogroup Y: ≥1:8 | 50.3 [43.0 to 57.5] | 50.0 [39.5 to 60.5]
  Serogroup Y: ≥1:128 | 27.7 [21.5 to 34.5] | 20.2 [12.6 to 29.8]
  Serogroup W 135: ≥1:8 | 20.0 [14.6 to 26.3] | 27.7 [18.9 to 37.8]
  Serogroup W 135: ≥1:128 | 12.8 [8.5 to 18.3] | 14.9 [8.4 to 23.7]

7. Primary Outcome: Percentage of Participants With Antibody Titers ≥1:8 and ≥1:128 Measured by rSBA Against Meningococcal Serogroups A, C, Y, and W 135 Following Vaccination With MenACYW Conjugate Vaccine or Menomune®
Description: Antibody titers against meningococcal serogroups A, C, Y, and W 135 were measured by rSBA assay method.
Time Frame: Day 30 (post-vaccination)
Population: Analysis was performed on PPAS population. Here, 'Overall number of participants analyzed' = participants evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: MenACYW Conjugate Vaccine | Group 2: Menomune® A/C/Y/W 135 Vaccine
Number analyzed (Participants) | 193 | 94
percentage of participants
  Serogroup A: ≥1:8 | 95.9 [92.0 to 98.2] | 94.7 [88.0 to 98.3]
  Serogroup A: ≥1:128 | 94.3 [90.0 to 97.1] | 89.4 [81.3 to 94.8]
  Serogroup C: ≥1:8 | 95.9 [92.0 to 98.2] | 87.2 [78.8 to 93.2]
  Serogroup C: ≥1:128 | 93.3 [88.8 to 96.4] | 77.7 [67.9 to 85.6]
  Serogroup Y: ≥1:8 | 97.4 [94.1 to 99.2] | 94.7 [88.0 to 98.3]
  Serogroup Y: ≥1:128 | 88.1 [82.7 to 92.3] | 73.4 [63.3 to 82.0]
  Serogroup W 135: ≥1:8 | 98.4 [95.5 to 99.7] | 94.7 [88.0 to 98.3]
  Serogroup W 135: ≥1:128 | 94.3 [90.0 to 97.1] | 79.8 [70.2 to 87.4]

8. Primary Outcome: Percentage of Participants With Vaccine Seroresponse Measured by rSBA Against Meningococcal Serogroups A, C, Y, and W 135 Following Vaccination With MenACYW Conjugate Vaccine or Menomune® Vaccine
Description: Vaccine seroresponse for serogroups A, C, Y, and W 135 was measured by rSBA assay method. Seroresponse was defined as post-vaccination rSBA titers ≥1:8 for participants with pre-vaccination rSBA titers <1:8, or at least a 4-fold increase in rSBA titers from pre- to post-vaccination for participants with pre-vaccination rSBA titers ≥1:8.
Time Frame: Day 30 (post-vaccination)
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: MenACYW Conjugate Vaccine | Group 2: Menomune® A/C/Y/W 135 Vaccine
Number analyzed (Participants) | 195 | 94
percentage of participants
  Serogroup A: number analyzed (Participants) | 193 | 93
  Serogroup A | 90.2 [85.1 to 94.0] | 89.2 [81.1 to 94.7]
  Serogroup C: number analyzed (Participants) | 193 | 94
  Serogroup C | 94.8 [90.7 to 97.5] | 86.2 [77.5 to 92.4]
  Serogroup Y: number analyzed (Participants) | 193 | 94
  Serogroup Y | 86.5 [80.9 to 91.0] | 75.5 [65.6 to 83.8]
  Serogroup W 135: number analyzed (Participants) | 193 | 94
  Serogroup W 135 | 95.3 [91.3 to 97.8] | 90.4 [82.6 to 95.5]

9. Primary Outcome: Geometric Mean Titers of Antibodies Against Meningococcal Serogroups A, C, Y, and W 135 Measured by rSBA Before Vaccination With MenACYW Conjugate Vaccine or Menomune® Vaccine
Description: GMTs of antibodies against meningococcal serogroups A, C, Y, and W 135 antibody titers were measured by rSBA assay method.
Time Frame: Day 0 (pre-vaccination)
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: titers (1/dilution)
Arm/Group | Group 1: MenACYW Conjugate Vaccine | Group 2: Menomune® A/C/Y/W 135 Vaccine
Number analyzed (Participants) | 195 | 94
titers (1/dilution)
  Serogroup A: number analyzed (Participants) | 195 | 93
  Serogroup A | 7.75 [5.65 to 10.6] | 7.32 [4.62 to 11.6]
  Serogroup C | 3.40 [2.76 to 4.18] | 2.93 [2.28 to 3.77]
  Serogroup Y | 15.3 [11.4 to 20.7] | 13.1 [8.63 to 19.9]
  Serogroup W 135 | 4.74 [3.68 to 6.12] | 6.05 [4.11 to 8.89]

10. Primary Outcome: Geometric Mean Titers of Antibodies Against Meningococcal Serogroups A, C, Y, and W 135 Measured by rSBA Following Vaccination With MenACYW Conjugate Vaccine or Menomune® Vaccine
Description: as for outcome 9
Time Frame: Day 30 (post-vaccination)
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: titers (1/dilution)
Arm/Group | Group 1: MenACYW Conjugate Vaccine | Group 2: Menomune® A/C/Y/W 135 Vaccine
Number analyzed (Participants) | 193 | 94
titers (1/dilution)
  Serogroup A | 1054 [825 to 1346] | 746 [501 to 1109]
  Serogroup C | 1559 [1140 to 2131] | 445 [255 to 776]
  Serogroup Y | 591 [464 to 753] | 260 [177 to 382]
  Serogroup W 135 | 910 [728 to 1136] | 493 [316 to 772]

11. Primary Outcome: Number of Participants With Immediate Unsolicited Adverse Events (AEs) After Vaccination
Description: An unsolicited AE was an observed AE that did not fulfill the conditions prelisted in the case report form (CRF) in terms of symptom and/or onset post-vaccination. Unsolicited AEs includes both serious and non-serious unsolicited AEs. A serious adverse event (SAE) was any untoward medical occurrence that at any dose resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect, or was an important medical event. All participants were observed for 30 minutes after vaccination, and any unsolicited AEs occurred during that time were recorded as immediate unsolicited AEs in the CRF.
Time Frame: Within 30 minutes after vaccination
Population: Analysis was performed on SafAS population which included participants who received at least one dose of the study or control vaccine and had safety data available.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: MenACYW Conjugate Vaccine | Group 2: Menomune® A/C/Y/W 135 Vaccine
Number analyzed (Participants) | 199 | 100
Participants | 0 | 0

12. Primary Outcome: Number of Participants With Solicited Injection Site Reactions and Systemic Reactions After Vaccination
Description: A solicited reaction (SR) was an adverse reaction (AR) observed and reported under the conditions (symptom and onset) prelisted in the CRF. Solicited injection site reactions included: pain, erythema, and swelling. Solicited systemic reactions included: fever, headache, malaise and, myalgia.
Time Frame: Within 7 days after vaccination
Population: Analysis was performed on SafAS population. Here, 'Number analyzed' = participants with available data for each specified category.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: MenACYW Conjugate Vaccine | Group 2: Menomune® A/C/Y/W 135 Vaccine
Number analyzed (Participants) | 199 | 100
Participants
  Pain | 61 | 32
  Erythema | 23 | 5
  Swelling: number analyzed (Participants) | 198 | 100
  Swelling | 15 | 2
  Fever: number analyzed (Participants) | 197 | 99
  Fever | 3 | 1
  Headache | 47 | 28
  Malaise | 44 | 15
  Myalgia | 70 | 26

13. Primary Outcome: Number of Participants With Unsolicited Adverse Events After Vaccination
Description: An unsolicited AE was an observed AE that does not fulfill the conditions prelisted in the CRF in terms of symptom and/or onset post-vaccination. Unsolicited AEs included both serious and non-serious unsolicited AEs. An SAE was any untoward medical occurrence that at any dose resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect, or was an important medical event. Non-serious AE (AE excluding SAE) which was significant and prevented daily activity was considered as Grade 3 unsolicited non-serious AE.
Time Frame: Within 30 days after vaccination
Population: Analysis was performed on the SafAS population.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: MenACYW Conjugate Vaccine | Group 2: Menomune® A/C/Y/W 135 Vaccine
Number analyzed (Participants) | 199 | 100
Participants
  Unsolicited AE | 41 | 17
  Unsolicited non-serious AE | 41 | 17
  Grade 3 unsolicited non-serious AE | 2 | 3

ADVERSE EVENTS:
Time Frame: Unsolicited AE data were collected from Day 0 up to Day 30 post-vaccination. The SRs were collected within 7 days post-vaccination. SAE information was collected throughout the trial (up to 30 days post-vaccination).
Description: A SR was an AE observed and reported under the conditions (symptom and onset) prelisted (i.e., solicited) in the CRF and considered to be related to vaccination. An unsolicited AE was an observed AE that did not fulfill the conditions prelisted in the CRF (i.e., solicited) in terms of symptom and/or onset post-vaccination. Analysis was performed on SafAS population.
Arm/Group | Group 1: MenACYW Conjugate Vaccine | Group 2: Menomune® A/C/Y/W 135 Vaccine
All-Cause Mortality (participants affected / at risk) | 0/199 | 0/100
Serious Adverse Events (participants affected / at risk) | 0/199 | 0/100
Other Adverse Events (participants affected / at risk) | 114/199 | 54/100
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: MenACYW Conjugate Vaccine (N=199) | Group 2: Menomune® A/C/Y/W 135 Vaccine (N=100)
Injection Site Erythema (General disorders) | 23 (23) | 5 (5)
Injection Site Pain (General disorders) | 61 (61) | 32 (32)
Injection Site Swelling (General disorders) | 15 (15) | 2 (2)
Malaise (General disorders) | 44 (44) | 15 (15)
Myalgia (Musculoskeletal and connective tissue disorders) | 70 (70) | 26 (26)
Headache (Nervous system disorders) | 47 (48) | 29 (30) — 1 Headache event which occurred 7 days post-vaccination was considered as an unsolicited AE.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable participant matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications.